CLINICAL TRIAL: NCT04372706
Title: Phase 1/2 Study of RTX-240 Monotherapy and in Combination With Pembrolizumab
Brief Title: RTX-240 Monotherapy and in Combination With Pembrolizumab
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated study during expansion on 11/30/22. RTX-240 was well-tolerated in multiple indications, combinations, and dose levels (69pts). No DLTs, related deaths or SAEs were reported. RTX-240 cleared circulation rapidly.
Sponsor: Rubius Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTX-240-01
Record Dates: First submitted 2020-04-23; First posted 2020-05-04 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Solid Tumor, AML Adult
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: RTX-240 Dose Escalation (Experimental): Phase 1: RTX-240 monotherapy dose escalation in Solid Tumors
  Interventions: Drug: RTX-240
- Part 2: RTX-240 Solid Tumor Expansion (Experimental): Phase 2: RTX-240 monotherapy dose expansion in Non-small Cell Lung Cancer (NSCLC), Renal Cell Carcinoma (RCC), and anal cancers
  Interventions: Drug: RTX-240
- Part 3: RTX-240 Dose Escalation (Experimental): Phase 1: RTX-240 monotherapy dose escalation in AML
  Interventions: Drug: RTX-240
- Part 4: RTX-240 Plus Pembrolizumab Dose Escalation (Experimental): Phase 1: RTX-240 dose escalation in combination with Pembrolizumab in Solid Tumors
  Interventions: Drug: RTX-240; Drug: Pembrolizumab

INTERVENTIONS:
Drug: RTX-240 — Engineered red cells co-expressing 4-1BBL and IL-15TP
Drug: Pembrolizumab — Humanized immunoglobulin G4 programmed death receptor-1 blocking antibody
  Arms: Part 4: RTX-240 Plus Pembrolizumab Dose Escalation

SUMMARY:
Open label, multicenter, multidose, first-in-human Phase 1/2 study of RTX-240 monotherapy or in combination of pembrolizumab for the treatment of patients with (1) relapsed/refractory R/R or locally advanced solid tumors (Phase 1/2) or (2) R/R Acute Myeloid Leukemia (AML) (Phase 1 only).

DETAILED DESCRIPTION:
This is a Phase 1/2, open label, multicenter, multidose, first-in-human (FIH) dose escalation and expansion study to determine the safety and tolerability, recommended phase 2 dose and optimal dosing interval, pharmacology, and antitumor activity of RTX-240 in adult patients with relapsed/refractory (R/R) or locally advanced solid tumors (Phase 1/2) or R/R acute myeloid leukemia (Phase 1 only), and RTX-240 in combination with pembrolizumab in adult patients with R/R or locally advanced solid tumors (Phase 1 only). RTX-240 is a cellular therapy that co-expresses 4-1BBL and IL-15TP, a fusion of IL-15 and IL-15 receptor alpha, with the goal of stimulating the innate and adaptive immune systems for the treatment of cancer. The study includes a monotherapy dose escalation phase (Phase 1) followed by an expansion phase (Phase 2) in specified tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to study procedures
* Patients ≥18 years with an ECOG 0 or 1 (Parts 1, 2 and 4) or 0-2 (Part 3).
* Relapsed/Refractory (R/R) or locally advanced, unresectable solid tumor for which no standard therapy exists (Parts 1, 2 and 4), or for which the patient is ineligible or has declined standard therapy or R/R, cytologically confirmed AML (Part 3).
* Disease must be measurable per Response Evaluation Criteria
* The shorter of 28 days or 5 half-lives must have elapsed since the completion of prior therapy, before initiation of study treatment.
* Adequate Organ Function and Blood Cell Counts (Parts 1, 2, and 4) as defined by the protocol:

  * GFR ≥ 50 mL/min/1.73,
  * AST and ALT ≤ 3 × the ULN and total bilirubin ≤ 1.5 × ULN, in the absence of cancer within the liver
  * Or AST and ALT ≤ 5 × ULN and total bilirubin ≤ 3 × ULN, in the setting of primary or metastatic liver tumors.
  * ANC ≥ 1 × 10^3/μL without myeloid growth factor support for at least one week prior to enrollment
  * Platelet count ≥ 75 × 10^3/μL
  * Hemoglobin should be ≥ 9 g/dL without red blood cell transfusion for at least one week
  * Patients must have LVEF ≥ 45%
* Patients enrolling into Part 2 of the study must be diagnosed with NSCLC, RCC, or anal cancers
* Patients enrolling into Part 4 must be diagnosed with NSCLC or RCC
* Patients enrolling into either Part 2 or 4 must have 2 or fewer prior treatment regimens. If patient received a prior PD-1/PD-L1-containing regimen, a prior response is required.

Exclusion Criteria:

* Primary central nervous system (CNS) malignancy or CNS involvement, unless asymptomatic, previously treated, and stable without steroids (Parts 1, 2 and 4) or known CNS leukemia (Part 3).
* Known hypersensitivity to any component of study treatment or excipients.
* Positive antibody screen using institution's standard type and screen test.
* Clinically significant, active and uncontrolled infection, including human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
* Clinically significant coagulopathy, uncontrolled hypertension or autoimmune hemolytic anemia
* Class III or IV cardiomyopathy per the New York Heart Association criteria
* Leukemic blast count ≥ 25 x 10^3/µL (Part 3)
* Concomitant conditions requiring active immunosuppression
* History of clinically significant Grade 3 or higher immune related Adverse Event (irAE)
* Prior malignancy within the past 3 years, with protocol specified exceptions
* History of severe hypersensitivity to a PD-1/PD-L1 blocking Ab unless previously rechallenged successfully (Part 4)
* Current noninfectious pneumonitis or a history of radiation pneumonitis or pneumonitis that required steroids, or Grade 2 or greater immune related pneumonitis, hepatitis, hypophysitis, or other endocrinopathy (Part 4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Safety Assessment: Measured by incidence of Treatment Emergent Adverse Events (TEAEs) | Up to 38 months
Dose limiting toxicities (DLTs) of study treatment as determined by incidence and severity of adverse events (AEs) | Up to 38 months

SECONDARY OUTCOMES:
PK of study treatment as measured by detection of the number of cells positive for both 4-1BBL and IL-15 using flow cytometry. | Assessed From the 1st dose of RTX-240 until 30 days after last of study treatment
Determination of the Immunogenicity of study treatment Measured by the incidence of antibodies to RTX-240 | Assessed From the 1st dose of RTX-240 until 30 days after last of study treatment
Anti-tumor activity of study treatment measured by clinical benefit rate (CBR) (% of patients who achieve CR, PR or stable disease [SD]) | Up to 38 months
Anti-tumor activity of study treatment measured by duration of response (DoR) | Up to 38 months
Anti-tumor activity of study treatment measured by progression free survival (PFS) | Up to 38 months
Anti-tumor activity of study treatment measured by overall survival (OS) | Up to 38 months
Anti-tumor activity of study treatment measured by time to response (TTR). | Up to 38 months
Anti-tumor activity of study treatment measured by time to progression (TTP) | Up to 38 months
Anti-Tumor activity of study treatment Measured by Objective Response Rate (ORR) | Up to 38 months
Proportion of AML patients with CR, CR with incomplete recovery (CRi), morphologic leukemia-free state, or PR | Up to 38 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of California San Diego, La Jolla, California
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - Sarah Cannon Research Institute/ Colorado Blood Cancer Institute, Denver, Colorado
  - Sylvester Comprehensive Cancer Center/UMHC, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Oregon Health & Sciences University - Knight Cancer Institute, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No